CLINICAL TRIAL: NCT05840653
Title: The Effect Of Posıtıve Psychotherapy-Based Hope Placement Program On The Level Of Determınatıon Of Hope And Lıve Goals In Indıvıduals Dıagnosed Wıth Multıple Sclerosıs
Brief Title: The Effect of Hope Placement Program on Dıagnosed Wıth MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Kubra Gulırmak, Research assistant in psychiatric nursing department, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: B.30.2.ODM.0.20.08/305
Record Dates: First submitted 2021-11-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; hope; life purpose; Psychiatric Nursing; positive psychotherapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This research is planned to be carried out as a Solomon Four-Group Experimental model. In the Solomon 2x2 designs, two of the four groups consisting of randomly assigned members by randomization constitute the experimental group and the other two constitute the control group. In the Solomon model, for statistical operations, pretesting is performed on two groups, one for the experimental group and the other for the control group, while the posttest process is performed on all four groups (Erkuş, 2011). The Solomon model is formed by using the pretest-posttest control group model and the posttest control group model together. In this way, the Solomon four-group experimental model is the strongest experimental model that preserves both internal and external validity (Karasar, 2011).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- experimental 1: Intervention group (Experimental): Experiment 1 group will first be given a pre-test, then a 5-week hope placement program will be applied. The final test will be administered after the program is completed.
  Interventions: Other: psychotherapeutic intervention
- experimental 2 group; Intervention group (Experimental): A 5-week hope placement program will be applied to the experimental 2 group without the pre-test application. After the program is completed, the final test will be administered.
  Interventions: Other: psychotherapeutic intervention
- control 1 group; not Intervention group (No Intervention): only the pre-test will be applied, other than that, no intervention will be applied in the 5-week period. Then the final test will be applied.
- control 2 group; not Intervention group (No Intervention): No intervention will be applied during the pre-test application and the 5-week period. then the final test will be administered.

INTERVENTIONS:
Other: psychotherapeutic intervention — The group that will receive 5-week positive psychotherapy-based hope placement psychoeducation
  Arms: experimental 1: Intervention group; experimental 2 group; Intervention group

SUMMARY:
Multiple Sclerosis (MS), causing damage to myelin sheath and axons; It is a chronic disease with diffuse demyelinating lesion of the Central Nervous System (CNS) that often affects young adults, progresses with attacks and remissions, and may bring about functional limitation, disability or decrease in quality of life. The fact that Multiple Sclerosis is chronic and irreversible, the uncertainty and destructiveness of the disease process affect individuals physically over time, but it can also cause many negative symptoms from a mental perspective. Studies have shown that MS disease; anxiety, depression, loss of life purpose, intense hopelessness and suicide. Life purpose has been defined as struggling to achieve one's goals and creating meaning against existential neurosis. Having a life purpose increases the subjective well-being, life satisfaction and hope level of individuals. According to the Turkish Language Association, hope, which is defined as "the feeling of trust arising from hope" and which indicates the feeling of having positive expectations for the future, positively affects mental health by giving people the feeling that they can cope with negative experiences that they may encounter in the future. Hopelessness, which is the opposite of hope, is a feeling that causes mental problems such as depression and suicide as well as negatively affecting the mental health of the individual and is a part of these clinical pictures. Setting a life purpose has positive effects on hope. While a purposeful life increases the level of hope in people, it reduces hopelessness and causes the person to live a more meaningful life. The decrease or loss of hope and the purpose of life can cause significant problems for people such as depression, addiction or suicide may occur in people who have lost their life purpose and hope. Positive psychotherapy (PPT), one of the psychosocial-based intervention methods, is a therapy method with a humanistic approach, the theoretical foundations of which were established by Pesesschkian in 1970. There are three basic principles of therapy: hope, balance and consultation. In Positive Psychotherapy, the symptoms and ailments in the person; It is positively reinterpreted, emphasizing real talents. Sharing the function of the existing symptom with the client increases the client's acceptance and hope for himself and his situation, which in turn activates the hope principle.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS), causing damage to myelin sheath and axons; It is a chronic disease with diffuse demyelinating lesion of the Central Nervous System (CNS) that often affects young adults, progresses with attacks and remissions, and may bring about functional limitation, disability or decrease in quality of life (Ertekin et al., 2012; Kuşçu et al., 2012; Milanlıoğlu et al., 2014; Daniel et al., 2018). Although the exact etiology of Multiple Sclerosis is not known, it is thought that many genetic and environmental factors may be effective (Veauthier, 2015; Brownlee et al., 2016). Multiple Sclerosis is more common in women than in men (Mitchell et al., 2019). An average of 50 thousand individuals diagnosed with Multiple Sclerosis inTurkey, It is reported that there are more than 2.5 million worldwide (Evans et al., 2013; Kalıncık et al., 2013; Akdemir et al. 2017; Mitchell et al., 2019). According to the data of the Turkish Statistical Institute (TUIK, 2018), MS ranks sixth among the causes of death with 4.1%, and ranks first among the diseases that cause disability. As it can be understood from the high rates of disability and death, it is a disease that imposes great burdens on a person's life (Gümüş, 2018; Tuncay, 2018; Öz & Öz, 2019).

The chronic and irreversible nature of Multiple Sclerosis disease, the uncertainty and destructiveness of the disease process affect individuals physically over time, and can also cause many negative symptoms in terms of mental health. Studies have shown that MS disease; anxiety, depression, loss of life purpose, intense hopelessness and suicide (1-2-3-4).

Life purpose has been defined as struggling to achieve one's goals and creating meaning against existential neurosis. Goals reflect the meaning, goals, and life tasks that are central to the psychological well-being perspective. Kasser and Ryan (1996) defined Life Goals as long-term goals that an individual hopes to achieve. Emmons (1992) defined life goals as situations that individuals try to achieve through cognitive and behavioral strategies. If individuals have set goals for themselves in different branches, it can be said that individuals have clarified their life goals. Nair (2003) states that life goals are also affected by previous positive or negative experiences. Looking at the literature, it is seen that life goals are handled with different classifications. For example, Pesesschkian's (1996) classification of life goals can be cited in the context of positive psychotherapy. Pesesschkian states that people set life goals in the areas of body (via senses), achievement (through career-mind), relationship (through traditions) and spirituality (via intuition). According to Pesesschkian (1996), people benefit from the resolution of conflicts in life by trying to achieve the goals they set in these four areas. Having a life purpose increases the subjective well-being, life satisfaction and hope level of individuals 5).

According to the Turkish Language Association, hope, which is defined as "the feeling of trust arising from hope" and which indicates the feeling of having positive expectations for the future, positively affects mental health by giving people the feeling that they can cope with negative experiences that they may encounter in the future. Hopelessness, which is the opposite of hope, is a feeling that causes mental problems such as depression and suicide as well as negatively affecting the mental health of the individual and is a part of these clinical pictures. Despair was also approved as a nursing diagnosis by the North American Nursing Diagnostic Association in 1986. Hope, which is important for human life, is perceived as a healing factor that empowers people to cope with momentary difficulties and overcome grief, and paves the way for finding meaning in life.

Setting a life purpose has positive effects on hope. While a purposeful life increases the level of hope in people, it reduces hopelessness and causes the person to live a more meaningful life. The decrease or loss of hope and the purpose of life can cause significant problems for people. Negative symptoms such as depression, addiction or suicide may occur in people who have lost their life purpose and hope. In such cases, in addition to the biological treatment methods applied to the person, the application of psychosocial-based interventions allows the symptoms to be resolved more easily.

The fact that Multiple Sclerosis is a chronic, uncertain, and exacerbating disease causes a decrease in the level of determination of life purpose from time to time or permanently, and hopelessness in the person. Therefore, focusing on problems such as "hopelessness and decreased life purpose" in individuals diagnosed with MS, teaching how to recognize and cope with symptoms, Positive psychotherapy (PPT), one of the psychosocial-based intervention methods, is a therapy method with a humanistic approach, the theoretical foundations of which were established by Pesesschkian. There are three basic principles of therapy: hope, balance and consultation. It is believed that real and existing things are not just conflicts and illnesses, but that there are innate abilities in every human being that accompany these conflicts and symptoms. In Positive Psychotherapy, the symptoms and ailments in the person; It is positively reinterpreted, emphasizing real talents. Sharing the function of the existing symptom with the client increases the client's acceptance and hope for himself and his situation, which in turn activates the hope principle (6). Again, starting from the principle of hope, there is this positive starting point, the principle of hope, related to each individual and situation at the center of PPT. Being talent and capacity oriented activates hope in the client and forms the basis of the healing process (7). The two important concepts mentioned, "hopelessness and life goals are among the main concepts of PPT. Therefore, it is thought that PPT-based psychoeducation will have a positive effect on situations such as hopelessness and low life purpose level.

When the international and national literature is examined, it is seen that the studies on PPT are limited. In addition, it has been found that most of the studies are related to depression, substance use disorder or university students (8-9-10-11-12). Studies using positive psychotherapy in patients diagnosed with Multiple Sclerosis are quite limited (13). In this respect, the research provides an opportunity for an up-to-date approach to the psychosocial problems of MS patients, and provides originality and importance in terms of contributing especially to the field of nursing and not having encountered a similar research topic in the literature.

ELIGIBILITY:
Inclusion Criteria

* Having been diagnosed with MS for at least 6 months,
* Not having a chronic disease diagnosis other than Multiple Sclerosis,
* Not having any diagnosed psychotic illness,
* Ability to read and write
* Being between the ages of 18-65,
* Not having a verbal or hearing disability that may affect communication,
* Owning a smart phone or computer,
* Ability to use the Internet, participate in online programs,
* Regular follow-up of psychoeducations,
* Participating in and completing all psychoeducational trainings,
* Filling the pretest and posttest questionnaires,
* Volunteering to participate in the study.
* Having an EDSS score of 6.5 and below. Exclusion Criteria
* Having a chronic disease other than Multiple Sclerosis,
* Not having any diagnosed psychotic illness,
* Having a verbal or hearing disability that may affect communication,
* Not having a smart phone or computer,
* Not having the ability to use the Internet or participate in online programs,
* Having an EDSS score of 6.5 and above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
experiment 1 and experiment 2 group level of determination of life purpose | 5 weeks
  In the experimental 1 and 2 groups, it is expected that there will be a significant increase in the total score of the life goals determination scale compared to the first test.
experiment 1 and experiment 2 group hopelessness is to decrease. | 5 weeks
  It is expected that there will be a significant decrease in the beck hopelessness scale total score in the experimental 1 and 2 groups compared to the first test.
control1 and control 2 group hopelessness is to decrease. | 5 weeks
  No change in life purpose and hopelessness level in Experiment 2 and Experiment 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: kübra gülırmak, MSc, Study Director — ONDOKUZ MAYIS UNİVERSITY; kübra gülırmak, msc, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- SAMSUN, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cope, T. (2010). The inherently integrative approach of Positive psychotherapy. The Journal of Psychotherapy Integration 20(2), 203-250.